CLINICAL TRIAL: NCT07406295
Title: Novel Respiratory Muscle Training for Improving Cerebrovascular Function and Immune Status in Adults With Obesity
Brief Title: Respiratory Muscle Training to Improve Cerebrovascular and Immune Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph Watso, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00006611
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Cerebrovascular Function; Immune Cells Activity
Keywords: Transcranial Doppler; Inspiratory Muscle Strength Training; Cerebrovascular Reactivity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: There is high intensity training group and low intensity (sham) group. Randomization is 2:1 for high to low intensity groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High intensity inspiratory muscle strength training (Active Comparator): Participants will perform high-resistance inspiratory muscle strength training on a daily basis for eight weeks using a handheld device that produces resistance that increases the effort of breathing in.
  Interventions: Device: High intensity inspiratory muscle strength training
- Low intensity inspiratory muscle strength training (Sham Comparator): Participants will perform very-low-resistance inspiratory muscle strength training on a daily basis for eight weeks using a handheld device that produces resistance that increases the effort of breathing in.
  Interventions: Device: Low intensity

INTERVENTIONS:
Device: High intensity inspiratory muscle strength training — This intervention will aim to increase inspiratory strength in adults with obesity to improve cerebrovascular function and immune status.
  Arms: High intensity inspiratory muscle strength training
Device: Low intensity — Very-low-resistance inspiratory muscle strength training
  Arms: Low intensity inspiratory muscle strength training

SUMMARY:
Millions of adults in America have too much body fat, resulting in obesity. Obesity is bad for health and causes disease. Obesity reduces brain health, which causes the brain to function worse. Also, a lack of exercise will make brain health worse. Most people feel they do not have time to exercise. There is a need for a quicker type of training that improves brain health.

Newly developed breathing exercises could be a time-efficient, cost-effective, and home-based practice to increase brain health. It is like weightlifting for your breathing muscles. These new breathing exercises have already been shown to increase heart health. Heart health is linked to brain health. If something helps the heart, it is likely to also help the brain. We do not know if breathing training can improve brain health in younger adults with obesity. We will use the same 8-week program shown to improve heart health. We will do testing before and after the breathing training. The first part of our study will determine if breathing exercises help brain health.

Obesity also causes inflammation. This is measured via blood but affects the entire body. It is thought to cause some of the negative outcomes of obesity. By lowering inflammation, it is likely to improve overall health. Breathing exercises may reduce inflammation, but more research is required. The second part of our study will determine whether breathing exercises help reduce inflammation.

This study will determine if we can improve brain health in adults with obesity. This could help 40% of American adults with obesity to live longer and healthier lives.

DETAILED DESCRIPTION:
Obesity, a growing global epidemic in America, is linked to cerebrovascular dysfunction and increases the risk of stroke, the nation's fourth leading cause of death. Cerebrovascular dysfunction is defined by impaired cerebrovascular reactivity and reduced cerebral autoregulation. Inspiratory muscle strength training (IMST) has proven to be a time-efficient, effective, low-cost, and highly feasible intervention for improving peripheral vascular function. Given the link between the peripheral vasculature and cerebrovasculature systems, it is highly plausible that IMST may improve cerebrovasculature function. There is emerging data showing that in adults with elevated blood pressure that IMST improves cerebrovascular function. Thus, the study team will examine whether 8 weeks of IMST improves cerebrovascular function in otherwise healthy young adults with obesity. Aim 1 will test the hypothesis that IMST will favorably increase cerebrovascular reactivity and improve cerebral autoregulation.

Obesity induced cerebrovascular dysfunction may be driven by chronic low-grade inflammation resulting from excessive sympathetic signaling. Additionally, inflammation is associated with reduced immune function. In adults with obesity, the systemic immune-inflammation index is elevated and positively associated with all-cause mortality. Emerging studies show IMST has the potential to reduce sympathetic activity and improve inflammation status. Aim 2 will test the hypothesis that IMST will reduce inflammation and improve immune function in otherwise healthy young adults with obesity.

We hypothesize that IMST will improve cerebrovascular reactivity and autoregulation, suggesting improved cerebrovascular health. Additionally, IMST will reduce systemic immune-inflammation index and improve immune function in otherwise healthy young adults with obesity.

This project explores the potential of IMST as a time-efficient and cost-effective intervention to improve cerebrovascular function and mitigate inflammation-related immune dysfunction in adults with obesity, potentially enhancing healthspan and lifespan. These findings could inform public health initiatives targeting approximately 40% of American adults with obesity, improving overall cerebrovascular function in the short term for adults with obesity, and reducing stroke incidence later in life.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal to 30 kg/m2
* Waist circumference greater or equal to 88 cm for females and greater than or equal to 102 cm for males

Exclusion Criteria:

* Not weight stable (<5% change in body mass over the past six months)
* Overt cardiovascular, neurological, renal, liver, and/or metabolic illness (e.g., diabetes mellitus)
* Current, or history of uncontrolled, Stage 2 hypertension (blood pressure >140 / 90 mmHg; anti-hypertensive medications are permitted)
* Diagnosed obstructive sleep apnea
* Previous bariatric surgery
* Diagnosis or signs (e.g., values below the lower limit of normal) of overt airway disease(s)
* Current or recent (regular use within the past 6 months) use of tobacco or nicotine products (e.g., cigarettes, vaping)
* Pregnant (self-reported and confirmed via urine pregnancy test), lactating (self-reported), or post-menopausal (self-reported) females
* Prisoners

Per the POWERbreathe® company:

* Patients who have undergone recent abdominal surgery and those with abdominal hernia.
* Asthma patients who have a very low symptom perception and suffer from frequent, severe exacerbations or with an abnormally low perception of dyspnea.
* If a patient is suffering from a ruptured eardrum or any other condition of the ear.
* Patients with marked elevated left ventricular end-diastolic volume and pressure.
* Patients with worsening heart failure signs and symptoms after training. If an individual is suffering from a cold, sinusitis or respiratory tract infection, it is advised that they do not use the POWERbreathe device.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in middle cerebral artery blood velocity reactivity to hypercapnia | Up to 9 weeks
  Middle cerebral artery blood velocity will be measured via transcranial Doppler ultrasound

SECONDARY OUTCOMES:
Change in immune cell androgenic sensitivity | Up to 9 weeks
  Isolate peripheral blood mononuclear cells and expose them to catecholamines to determine concentration of cAMP production.
Change in dynamic cerebral autoregulation phase | Up to 9 weeks
  Calculated from middle cerebral artery blood velocity signal using transfer function analysis
Change in total resting brain blood flow | Up to 9 weeks
  Total brain blood flow measured in the internal carotid and vertebral arteries at rest via ultrasound
Change in dynamic cerebral autoregulation gain | Up to 9 weeks
  Calculated from middle cerebral artery blood velocity signal using transfer function analysis
Middle cerebral artery blood velocity pulsatility index | Up to 9 weeks
  Calculated from middle cerebral artery blood velocity signal

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Watso, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided